CLINICAL TRIAL: NCT06752694
Title: Ruxolitinib Based GVHD Prophylaxis Regimen for Older Adults Receiving Non-ATG Containing Non-Myeloablative Hematopoietic Cell Transplantation for Acquired Aplastic Anemia
Brief Title: Ruxolitinib Based GVHD Prophylaxis Regimen Before, During, and After Hematopoietic Cell Transplantation in Older Adult Patients With Acquired Aplastic Anemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1124040; NCI-2024-06524 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20575 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Specimen Handling; Biopsy; Bone Marrow Transplantation; Blood Specimen Collection; Cyclosporine; Cyclosporins; fludarabine; Granulocyte Colony-Stimulating Factor; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; ruxolitinib; Sirolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (conditioning, transplant, GVHD prophylaxis) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Transplantation; Procedure: Computed Tomography; Drug: Cyclosporine; Drug: Fludarabine; Drug: Granulocyte Colony-Stimulating Factor; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Ruxolitinib; Drug: Sirolimus; Radiation: Total-Body Irradiation; Procedure: Multigated Acquisition Scan; Procedure: Echocardiography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Bone Marrow Transplantation — Undergo bone marrow transplant
  Other Names: Blood and Bone Marrow Transplant; BMT; Bone Marrow; Bone Marrow Grafting; Bone Marrow Transplant; Marrow Transplantation
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; CyA; Cyclosporin; Cyclosporin A; Cyclosporine Modified; Gengraf; Neoral; OL 27-400; Sandimmune; SangCya
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Granulocyte Colony-Stimulating Factor — Given SC
  Other Names: Colony Stimulating Factor 3; Colony-Stimulating Factor (Granulocyte); Colony-Stimulating Factor 3; CSF3; G CSF; G-CSF; GCSF; Granulocyte Colony Stimulating Factor; Pluripoietin
Drug: Mycophenolate Mofetil — Given PO
  Other Names: CellCept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC transplantation
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Drug: Ruxolitinib — Given PO
  Other Names: INCB 018424; INCB-018424; INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424
Drug: Sirolimus — Given PO
  Other Names: AY 22989; AY-22989; AY22989; RAPA; Rapamune; Rapamycin; SILA 9268A; SILA-9268A; SILA9268A; WY 090217; WY-090217; WY090217
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body; Whole Body Irradiation; Whole-Body Irradiation
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: MUGA; MUGA Scan; Radionuclide ventriculography
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC

SUMMARY:
This phase II trial tests how well a ruxolitinib-based graft versus host disease (GVHD) prevention (prophylaxis) regimen works before, during, and after bone marrow/stem cell transplantation (hematopoietic cell transplantation [HCT]) in patients with acquired aplastic anemia. Acquired aplastic anemia (AA) is a condition in which the bone marrow is unable to produce blood cells. Affected patients typically present with infections due to abnormally low number of neutrophils, bleeding due to low platelet count, and/or fatigue due to a lower-than-normal number of red blood cells (anemia). Its incidence varies with age, occurring most frequently in patients aged 2-5 years, 20-25 years, and 55 years and older. Treatment of AA includes either immunosuppressive therapy (IST) or bone marrow/stem cell transplantation (HCT) with first-line therapy in younger adults often being HCT, while adults over 40 still frequently trial IST first due to the morbidity and mortality concerns with HCT. GVHD is a common complication after donor stem cell transplantation, resulting from donor immune cells recognizing recipients' cells and attacking them. Ruxolitinib, a drug in a class of oral medications called JAK inhibitors has been approved for the treatment of acute and chronic GVHD. It has also been shown to decrease GVHD when used in the prevention setting in patients with myelofibrosis. The current study aims to assess whether adding ruxolitinib to a standard GVHD prevention regimen may reduce the risk of Grade II-IV acute and chronic GVHD after bone marrow/stem cell transplantation in older patients with acquired aplastic anemia.

DETAILED DESCRIPTION:
OUTLINE:

CONDITIONING REGIMEN: Patients receive fludarabine intravenously (IV) over 30 minutes once daily (QD) on days -4, -3, and -2 and undergo total body irradiation (TBI) in one or two fractions on day -1.

TRANSPLANT: Patients undergo peripheral blood stem cell (PBSC) or bone marrow transplant on day 0.

GVHD PROPHYLAXIS: Cyclosporine, Sirolimus, mycophenolate mofetil (MMF), Ruxolitinib

HUMAN LEUKOCYTE ANTIGEN (HLA)-MATCHED: Patients receive cyclosporine orally (PO) every 12 hours (Q12H) on days -3 to 96 with taper beginning on day 97 until day 180 (until day 150 for patients with unrelated donors), ruxolitinib PO twice daily (BID) or QD on day -5 to 365 and mycophenolate mofetil (MMF) PO 4-6 hours after transplant and then every 8 hours (Q8H) until day 29, then reduced to Q12H on days 30-40. Patients with unrelated donors also receive sirolimus PO QD on days -3 to 150 with taper beginning on day 151 until day 180. Patients also begin granulocyte colony-stimulating factor (G-CSF) subcutaneously (SC) on day 1 to continue until absolute neutrophil count (ANC) > 1000/mm^3 x 3 days. Patients also undergo multi-gated acquisition scan (MUGA)/echocardiogram (ECHO) and computed tomography (CT) during screening, as well as collection of blood samples and bone marrow aspiration and biopsy throughout the study.

HLA-MISMATCHED: Patients receive cyclosporine PO Q12 on days -3 to 150 with taper beginning on day 151 until day 180, sirolimus PO QD on days -3 to 180 with taper beginning on day 181 until day 365, ruxolitinib PO BID or QD on day -5 to 365, and MMF PO 4-6 hours after transplant and then Q8 until day 29, then reduced to Q12H on days 30-40. Patients also begin G-CSF SC on day 1 to continue until ANC > 1000/mm^3 x 3 days.

Patients also undergo MUGA/ECHO and CT during screening, as well as collection of blood samples and bone marrow aspiration and biopsy throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years or ages 18 - 40 years with Hematopoietic Cell Transplantation - Specific Comorbidity Index (HCT-CI) score > 3 necessitating a low intensity transplant or determined inability to tolerate antithymocyte globulin (ATG)
* Diagnosis of severe acquired aplastic anemia defined as a bone marrow hypoplasia (< 25% or 25-50% with < 30% residual hematopoietic cells) shown by a biopsy and at least two of the three following criteria: absolute neutrophil count (ANC) < 0.5×10^9/L, platelets < 20×10^9/L, or absolute reticulocytes < 40×10^9/L or
* Non-severe acquired aplastic anemia defined as a hypocellular marrow and transfusion dependent (red cells and/or platelets)
* Does not meet World Health Organization (WHO) criteria for myelodysplastic syndrome (MDS)
* Ability to understand and the willingness to sign a written informed consent document
* Patient must be a potential hematopoietic stem cell transplant candidate as assessed by the consenting physician
* Karnofsky ≥ 70
* Calculated creatinine clearance using the Cockcroft-Gault formula or 24 hr urine creatinine clearance must be > 60 ml/min
* Total serum bilirubin must be < 2 mg/dL unless the elevation is thought to be due to Gilbert's disease or hemolysis
* Transaminases must be < 3x the upper limit of normal
* Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension. Patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, hepatic encephalopathy, or correctable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3mg/dL, and symptomatic biliary disease will be excluded
* Diffusing capacity for carbon monoxide (DLCO) corrected > 60% normal
* May not be on supplemental oxygen
* Left ventricular ejection fraction > 40% OR shortening fraction > 26%
* Patients may have received prior treatment for their AA but they are NOT required to have received immune suppression prior to consideration for transplant

Exclusion Criteria:

* Contraindication to receiving ruxolitinib including: patients who have known hypersensitivity to JAK inhibitors and excipients
* Patients with history of myocardial infarction (MI), cerebrovascular accident (CVA) or unprovoked pulmonary embolism (PE)/deep vein thrombosis (DVT) in past 6 months
* History of prior allogeneic transplant
* Active or recent infection without infectious disease (ID) consult and approval
* History of untreated tuberculosis (TB)
* History of HIV infection
* Pregnant or breastfeeding
* History of prior malignancy with > 20% risk of recurrence in the next 5 years
* Patients without an HLA-identical sibling donor, 10 of 10 HLA-matched or 9 of 10 mismatched unrelated donor that meet transplant criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grades II-IV acute graft-versus-host disease (GVHD) | At day 100
  Will be estimated as simple proportions and informally compared to the historical controls at Fred Hutch. (i.e., estimates presented descriptively, but no formal statistical comparisons will be made).

SECONDARY OUTCOMES:
Incidence of grade III-IV acute GVHD | At day 100
  Will be estimated as simple proportions and informally compared to the historical controls at Fred Hutch. (i.e., estimates presented descriptively, but no formal statistical comparisons will be made).
Incidence of chronic GVHD | At 1 year
  Will be estimated as simple proportions and informally compared to the historical controls at Fred Hutch. (i.e., estimates presented descriptively, but no formal statistical comparisons will be made).
Incidence of primary graft failure | At 2 years
  Will be defined as absence of 3 consecutive days with neutrophils ≥ 500/ul combined with host CD3 peripheral blood chimerism ≥ 50% at day 42; absence of 3 consecutive days with neutrophils ≥ 500/ul under any circumstances at day 55; death after day 28 with neutrophil count <100/ul without any evidence of engraftment (< 5% donor CD3) and; primary autologous count recovery with < 5% donor CD3 peripheral blood chimerism at count recovery and without relapse.
Nonrelapse mortality | At day 100
  Kaplan-Meier curve will be generated with point estimates and 95% confidence intervals, and Log-rank test will be conducted.
Overall survival | At 1 year
  Kaplan-Meier curve will be generated with point estimates and 95% confidence intervals, and Log-rank test will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B. Salit, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No